CLINICAL TRIAL: NCT06526975
Title: Study of Different Exercise Doses Through Digital Gamification in Older Adults
Brief Title: Study of Different Exercise Doses Through Videogames in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBA-01
Record Dates: First submitted 2024-07-15; First posted 2024-07-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Older Adult

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gamification 10-20' (Experimental): This group will perform between 10 and 20 minutes of exercise through different videogames.
  Interventions: Other: Gamification exercise through a videogame
- Gamification 20-30' (Experimental): This group will perform between 20 and 30 minutes of exercise through different videogames.
  Interventions: Other: Gamification exercise through a videogame

INTERVENTIONS:
Other: Gamification exercise through a videogame — Different exercises will be performed through a videogame.

SUMMARY:
The objective of this clinical trial is to assess the feasibility of applying different gamified exercises doses in older adults. It will also learn from possible adverse effects of the intervention.

The main questions this clinical trial aims to answer are:

* Are there any differences between heart rate, perceived exertion and enjoyment between groups?
* Are there any adverse effects? What is the magnitude of these adverse effects?
* Are there any correlations between gamification time and the occurrence of adverse effects?

DETAILED DESCRIPTION:
A randomised clinical trial will be conducted in which the use of exercise doses between 10 and 30 will be tested. Participants will be recruited from Nueva Esperanza nursing home, Fuensalida, Toledo. The study will be conducted according to the CONSORT statement for clinical, crossover and parallel trials.

The study will have a total of two experimental groups, with different intervention times, between 10 and 30 minutes, respectively, using a mobile application. The intervention will consist of performing exercise in pairs in a single bout during the mentioned times.

ELIGIBILITY:
Inclusion Criteria:

* subjects over 60 years of age
* score equal to or greater than 20 on the Mini Mental cognitive test
* Subjects that present the ability to stand without the use of technical aids or with the technical assistance of a device used for walking.

Exclusion Criteria:

* severe visual impairment
* medical contraindication for physical activity
* pathology or problem that could prevent the test from being carried out.

Ages: 60 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate | Heart rate is measured thourought the intervention, once the intervention is finished (10 to 30 minutes) recording of heart rate will stop.
  Heart rate will be measured using polar H10
Rate of perceived exertion | RPE will be measured at half time and once the intervention is finished for both groups.
  Rate of perceived exertion will be measured using Borg (RPE 6-20). Higher values indicate higher levels of perceived exertion
Exercise satisfaction | It will be measured on the same day intervention finishes, up to 5 hours post-intervention.
  It will be measured using Physical Activity Enjoyment Scale (PACES). Higher values indicate higher percieved satisfaction/ enjoyment
Adverse effects | 24 and 48 hours post-intervention
  It will be measured using Hooper and Mackinnon wellness questionnaire. Higher values indicate worse perceived effects.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Nueva Esperanza Nursing Home, Fuensalida, Toledo
  - Universidad de Castilla La Mancha, Toledo, Toledo

IPD SHARING:
Plan to Share IPD: Undecided
Data will be provided to other researchers if asked to the principal investigator